CLINICAL TRIAL: NCT00508976
Title: Evaluation of Aerosolized Bupivacaine Versus Pre-incision Lidocaine Versus Instilled Liquid Bupivacaine Versus Post-operative Bupivacaine Injection for Optimization of Post-operative Pain Control in Laparoscopic Bariatric Surgical Patients
Brief Title: Clinical Proposal for the Comparison of Intraperitoneal Anesthetic to Injected Local Anesthetic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pinnacle Health System (Other)
Responsible Party: Principal Investigator, Troy Moritz, D.O., Troy Moritz DO, Pinnacle Health System
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: PHH#07-005
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Pain, Postoperative; Morbid Obesity
Keywords: bupivacaine; marcaine; lidocaine; normal saline; narcotics; analog pain scale; postoperative pain; preemptive; aerosolization; streamed
MeSH Terms: conditions — Pain, Postoperative; Obesity, Morbid | interventions — Bupivacaine; Saline Solution; Aerosolized Particles and Droplets; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 3 (Experimental)
  Interventions: Drug: Streamed bupivacaine versus streamed normal saline
- 2 (Experimental)
  Interventions: Drug: Injected lidocaine pre-incision vs saline pre-incision
- 4 (Experimental)
  Interventions: Drug: Aerosolized bupivacaine versus aerosolized saline
- 1 (Active Comparator)
  Interventions: Drug: Injected bupivacaine post-operatively

INTERVENTIONS:
Drug: Injected bupivacaine post-operatively — Patients will receive 30 ml of 0.9% normal saline divided equally and injected prior to port site incision, then 10ml of 0.9% normal saline streamed via port directed at operative field, then 10ml of 0.9% normal saline aerosolized into the coelomic cavity prior to deflation, and our current standard of care, which is 30ml of 0.5% bupivacaine, divided equally between the five port-sites, injected at the end of the operation.
  Other Names: bupivacaine
  Arms: 1
Drug: Streamed bupivacaine versus streamed normal saline — Patients will receive 30ml of 0.9% normal saline divided equally and injected prior to port site incisions, then 10ml of 0.5% bupivacaine streamed via port directed at operative field, then 10ml of 0.9% normal saline aerosolized into the coelomic cavity prior to deflation and our current standard of care, which is 30ml of 0.5% bupivacaine, divided equally between the five port-sites, injected at the end of the operation.
  Other Names: bupivacaine; marcaine; normal saline
  Arms: 3
Drug: Aerosolized bupivacaine versus aerosolized saline — Patients will receive 30 ml of 0.9% normal saline divided equally and injected prior to port site incision, then 10ml of 0.9% normal saline streamed via port directed at operative field, then 10ml of 0.5% bupivacaine aerosolized into coelomic cavity prior to deflation and our current standard of care, which is 30ml of 0.5% bupivacaine, divided equally between the five port-sites, injected at the end of the operation.
  Other Names: bupivacaine; marcaine; normal saline; aerosolized
  Arms: 4
Drug: Injected lidocaine pre-incision vs saline pre-incision — Patients will receive 30ml of 1% lidocaine divided equally and injected prior to port site incisions, then 10ml of 0.9% normal saline streamed via port directed at operative field, then 10ml of 0.9% normal saline aerosolized into the coelomic cavity prior to deflation and our current standard of care, which is 30ml of 0.5% bupivacaine, divided equally between the five port-sites, injected at the end of the operation.
  Other Names: lidocaine; normal saline; pre-emptive
  Arms: 2

SUMMARY:
The purpose of this study is to determine if pre-incisional lidocaine injection, instilled liquid bupivacaine, intra-abdominal aerosolized bupivacaine, or post-operative bupivacaine injection is superior in post-operative pain control in laparoscopic bariatric surgical patients.

DETAILED DESCRIPTION:
The research objective is to compare our standard post-operative port site injection of 0.5% bupivacaine against pre-incisional port site injection of 1% lidocaine against the instillation of streamed bupivacaine 0.5% against the instillation of aerosolized 0.5% bupivacaine as it relates to post-operative analgesia usage and pain scale scores. The null hypothesis will be that there is no difference between the four arms of the study in regards to pain score and analgesia usage.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between 18 and 65 years of age.
2. Patients undergoing elective bariatric surgery.

Exclusion Criteria:

1. Patients allergic to bupivacaine or any other local anesthetics (amides & esters).
2. Patients who have used opiates or opiods within 15 days prior to surgery.
3. Patients converted to open gastric bypass.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Measure of reduction in post-operative pain and narcotics usage. | First 3 days post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Troy A Moritz, DO, Principal Investigator — Pinnacle Health; Community General Osteopathic Hospital
Locations (1):
- Pinnacle Health; Community General Osteopathic Hospital, Harrisburg, Pennsylvania, United States

REFERENCES:
- [Background] Aida S, Baba H, Yamakura T, Taga K, Fukuda S, Shimoji K. The effectiveness of preemptive analgesia varies according to the type of surgery: a randomized, double-blind study. Anesth Analg. 1999 Sep;89(3):711-6. doi: 10.1097/00000539-199909000-00034. PMID 10475311
- [Background] Alkhamesi NA, Peck DH, Lomax D, Darzi AW. Intraperitoneal aerosolization of bupivacaine reduces postoperative pain in laparoscopic surgery: a randomized prospective controlled double-blinded clinical trial. Surg Endosc. 2007 Apr;21(4):602-6. doi: 10.1007/s00464-006-9087-6. Epub 2006 Dec 16. PMID 17180268
- [Background] Barczynski M, Konturek A, Herman RM. Superiority of preemptive analgesia with intraperitoneal instillation of bupivacaine before rather than after the creation of pneumoperitoneum for laparoscopic cholecystectomy: a randomized, double-blind, placebo-controlled study. Surg Endosc. 2006 Jul;20(7):1088-93. doi: 10.1007/s00464-005-0458-1. Epub 2006 May 13. PMID 16703434
- [Background] Chou YJ, Ou YC, Lan KC, Jawan B, Chang SY, Kung FT. Preemptive analgesia installation during gynecologic laparoscopy: a randomized trial. J Minim Invasive Gynecol. 2005 Jul-Aug;12(4):330-5. doi: 10.1016/j.jmig.2005.05.005. PMID 16036193
- [Background] Einarsson JI, Sun J, Orav J, Young AE. Local analgesia in laparoscopy: a randomized trial. Obstet Gynecol. 2004 Dec;104(6):1335-9. doi: 10.1097/01.AOG.0000146283.90934.fd. PMID 15572499
- [Background] Fletcher D, Kayser V, Guilbaud G. Influence of timing of administration on the analgesic effect of bupivacaine infiltration in carrageenin-injected rats. Anesthesiology. 1996 May;84(5):1129-37. doi: 10.1097/00000542-199605000-00015. PMID 8624007
- [Background] Huang SJ, Wang JJ, Ho ST, Liu HS, Liaw WJ, Li MJ, Liu YH. The preemptive effect of pre-incisional bupivacaine infiltration on postoperative analgesia following lower abdominal surgery under epidural anesthesia. Acta Anaesthesiol Sin. 1997 Jun;35(2):97-102. PMID 9293650
- [Background] Ke RW, Portera SG, Bagous W, Lincoln SR. A randomized, double-blinded trial of preemptive analgesia in laparoscopy. Obstet Gynecol. 1998 Dec;92(6):972-5. doi: 10.1016/s0029-7844(98)00303-2. PMID 9840560
- [Background] Kundu S, Achar S. Principles of office anesthesia: part II. Topical anesthesia. Am Fam Physician. 2002 Jul 1;66(1):99-102. PMID 12126037
- [Background] Lam KW, Pun TC, Ng EH, Wong KS. Efficacy of preemptive analgesia for wound pain after laparoscopic operations in infertile women: a randomised, double-blind and placebo control study. BJOG. 2004 Apr;111(4):340-4. doi: 10.1111/j.1471-0528.2004.00083.x. PMID 15008770
- [Background] Lohsiriwat V, Lert-akyamanee N, Rushatamukayanunt W. Efficacy of pre-incisional bupivacaine infiltration on postoperative pain relief after appendectomy: prospective double-blind randomized trial. World J Surg. 2004 Oct;28(10):947-50. doi: 10.1007/s00268-004-7471-8. Epub 2004 Sep 29. PMID 15573244
- [Background] Jiranantarat V, Rushatamukayanunt W, Lert-akyamanee N, Sirijearanai R, Piromrat I, Suwannanonda P, Muangkasem J. Analgesic effect of intraperitoneal instillation of bupivacaine for postoperative laparoscopic cholecystectomy. J Med Assoc Thai. 2002 Sep;85 Suppl 3:S897-903. PMID 12452227
- [Background] Maestroni U, Sortini D, Devito C, Pour Morad Kohan Brunaldi F, Anania G, Pavanelli L, Pasqualucci A, Donini A. A new method of preemptive analgesia in laparoscopic cholecystectomy. Surg Endosc. 2002 Sep;16(9):1336-40. doi: 10.1007/s00464-001-9181-8. Epub 2002 May 7. PMID 11988800
- [Background] Mixter CG 3rd, Hackett TR. Preemptive analgesia in the laparoscopic patient. Surg Endosc. 1997 Apr;11(4):351-3. doi: 10.1007/s004649900361. PMID 9094275
- [Background] Moiniche S, Kehlet H, Dahl JB. A qualitative and quantitative systematic review of preemptive analgesia for postoperative pain relief: the role of timing of analgesia. Anesthesiology. 2002 Mar;96(3):725-41. doi: 10.1097/00000542-200203000-00032. No abstract available. PMID 11873051
- [Background] Mouton WG, Bessell JR, Otten KT, Maddern GJ. Pain after laparoscopy. Surg Endosc. 1999 May;13(5):445-8. doi: 10.1007/s004649901011. PMID 10227938
- [Background] Mouton WG, Bessell JR, Pfitzner J, Dymock RB, Brealey J, Maddern GJ. A randomized controlled trial to determine the effects of humidified carbon dioxide insufflation during thoracoscopy. Surg Endosc. 1999 Apr;13(4):382-5. doi: 10.1007/s004649900994. PMID 10094752
- [Background] Mouton WG, Bessell JR, Millard SH, Baxter PS, Maddern GJ. A randomized controlled trial assessing the benefit of humidified insufflation gas during laparoscopic surgery. Surg Endosc. 1999 Feb;13(2):106-8. doi: 10.1007/s004649900915. PMID 9918607
- [Background] Ong CK, Lirk P, Seymour RA, Jenkins BJ. The efficacy of preemptive analgesia for acute postoperative pain management: a meta-analysis. Anesth Analg. 2005 Mar;100(3):757-773. doi: 10.1213/01.ANE.0000144428.98767.0E. PMID 15728066